CLINICAL TRIAL: NCT01831700
Title: A Randomized, Open Label, Balanced, Two-Treatment, Two-Period, Two-Sequence, Single Dose, Crossover, Comparative Bioavailability Study of Lisinopril and Hydrochlorothiazide Tablets (20+25) mg of M/s Ipca Laboratories Ltd., India With Zestoretic® 20/25 Lisinopril/Hydrochlorothiazide Tablets of M/s AstraZeneca Pharmaceuticals LP, USA in Normal, Healthy, Adult, Human Subjects Under Fasting Condition
Brief Title: Bioequivalence Study of Lisinopril and Hydrochlorothiazide Tablets (20+25) mg Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IPCA Laboratories Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Ipca/ARL/10/386
Record Dates: First submitted 2013-04-05; First posted 2013-04-15 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting | interventions — Lisinopril; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lisinopril and Hydrochlorothiazide Tablets (20+25) mg (Experimental): Lisinopril and Hydrochlorothiazide Tablets (20+25) mg of M/s Ipca Laboratories Ltd., India
  Interventions: Drug: Lisinopril and Hydrochlorothiazide Tablets (20+25) mg; Drug: Zestoretic® 20/25 lisinopril/hydrochlorothiazide Tablets
- Zestoretic® 20/25 lisinopril/hydrochlorothiazide Tablets (Active Comparator): Zestoretic® 20/25 lisinopril/hydrochlorothiazide Tablets of M/s AstraZeneca Pharmaceuticals LP, USA
  Interventions: Drug: Lisinopril and Hydrochlorothiazide Tablets (20+25) mg; Drug: Zestoretic® 20/25 lisinopril/hydrochlorothiazide Tablets

INTERVENTIONS:
Drug: Lisinopril and Hydrochlorothiazide Tablets (20+25) mg — Lisinopril and Hydrochlorothiazide (20+25) mg Tablets once a day
  Other Names: Test product
Drug: Zestoretic® 20/25 lisinopril/hydrochlorothiazide Tablets — Zestoretic® 20/25 lisinopril/hydrochlorothiazide Tablets once a day
  Other Names: Reference product

SUMMARY:
This is a randomized, open Label, balanced, two-treatment, two-period, two-sequence, single dose, cross over pivotal study. The purpose of this study is to assess the bioequivalence between Test Product and the corresponding Reference Product under fasting condition in normal, healthy, adult, human subjects.

DETAILED DESCRIPTION:
Objective of this pivotal study was to assess the bioequivalence between Test Product: Lisinopril and Hydrochlorothiazide Tablets (20+25) mg of M/s Ipca Laboratories Ltd., India and the corresponding Reference Product: Zestoretic® 20/25 lisinopril/hydrochlorothiazide Tablets of M/s AstraZeneca Pharmaceuticals LP, USA under fasting condition in normal, healthy, adult, human subjects in a randomized crossover study.

The study was conducted with 48 healthy adult subjects. In each study period, a single Lisinopril and Hydrochlorothiazide Tablets (20+25) mg of either test or reference was administered to the subjects as per the randomization schedule in each study period with about 240 mL of water at ambient temperature in sitting position.

The duration of clinical phase was 12 days, including the washout period of 7 days between each study period.

ELIGIBILITY:
Inclusion Criteria:

1. Male and non-pregnant female human subjects, age in the range of 18 - 45 years (both inclusive).
2. Subject willing to give written informed consent.
3. Body weight within ± 15% of ideal weight as related to height and body frame according to Life Insurance Corporation (LIC) Chart.
4. Subjects with normal findings as determined by baseline history, physical examination and vital signs (blood pressure, pulse rate, respiration rate and oral temperature).
5. Subjects with clinically acceptable findings as determined by haemogram, biochemistry including serum electrolytes test, serology (HIV, Hepatitis B and Hepatitis C), urinalysis, 12 lead ECG and chest X-ray (chest X-ray if taken).
6. Willingness to follow the protocol requirements as evidenced by written informed consent.
7. Confirming and agreeing to, not using any prescription and over the counter medications including vitamins and minerals for 14 days prior to study & during the course of the study.
8. No history of drug abuse in the past one year.
9. Non-smokers and Non-alcoholics.
10. For female subject:

    * Was child bearing potential practicing acceptable method of birth control for the duration of the study as judged by Investigator such as Condom, Foams, Jellies, Diaphragm , Intrauterine device and Abstinence. OR
    * Was surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy has been performed on the subject).

Exclusion Criteria:

1. Known history of hypersensitivity to Lisinopril and Hydrochlorothiazide, other sulfonamide-derived drugs or related drugs.
2. Requiring medication for any ailment having enzyme-modifying activity in the previous 28 days, prior to dosing day.
3. Any medical or surgical conditions, which might significantly interfere with the functioning of gastrointestinal tract, blood-forming organs etc.
4. History of cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic, hematological, gastrointestinal, endocrine, immunological or psychiatric diseases and bleeding tendency.
5. Participation in a clinical drug study or bioequivalence study within 90 days prior to present study.
6. History of malignancy or other serious diseases.
7. Refusal to abstain from food from at least ten (10.00) hours prior to study drug administration until at least four (04.00) hours post-dose, in each study period.
8. Any contraindication to blood sampling or difficulty in accessibility of veins.
9. Refusal to abstain from fluid from at least 01.00 hour prior to study drug administration until at least 01.00 hour post-dose, in each study period except about 240 mL of water given during administration of study drug.
10. Refusal to avoid the use of xanthine-containing food or beverages (chocolates, tea, coffee or cola drinks) or fruit juice/grapefruit juice and any alcoholic products for 48.00 hours prior to dosing until the last blood sample collection of last study period.
11. Blood donation within 90 days prior to the commencement of the study.
12. Subjects with positive HIV tests or Hepatitis-B or Hepatitis-C tests.
13. Found positive in breath alcohol test done before check-in for each study period.
14. Found positive in urine test for drug abuse done before check-in for each study period.
15. Refusal to abstain from consumption of tobacco products 24.00 hours prior to dosing until the last blood sample collection of last study period.
16. History of problem in swallowing tablet(s).
17. Female subject, demonstrating positive urine pregnancy test at the time of screening.
18. Female subject, demonstrating positive Serum (ß) Beta- hCG (Human Chorionic Gonadotropin) test before check-in for each study period.
19. Female subject, currently breast feeding or lactating.
20. Female subjects not willing to use acceptable method of contraception from the date of screening until the completion of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence is based on Cmax and AUC parameters. | 1 Months
  Sampling Hours: Pre-dose and at 00.50, 01.00, 01.50, 02.00, 02.50, 03.00, 03.50, 04.00, 04.50, 05.00, 05.50, 06.00, 06.50, 07.00, 07.50, 08.00, 09.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00 and 72.00 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Tarang Girishbhai Shah, M. D. (Pharmacology), Principal Investigator — Accutest Research Lab (I) Pvt. Ltd.
Locations (1):
- Accutest Research Lab (I) Pvt. Ltd., Ahmedabad, Gujarat, India